CLINICAL TRIAL: NCT02330705
Title: Timing of Human Chorionic Gonadotropin Administration in Intrauterine Insemination Cycles
Brief Title: Timing of HCG Administration in IUI Cycles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Ibrahem Eid (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ibrahem Eid, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MIE3
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Infertility
Keywords: Intrauterine insemination; IUI; HCG
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): IUI at time of HCG
  Interventions: Drug: HCG
- Group B (Active Comparator): IUI 12 hours after HCG
  Interventions: Drug: HCG
- Group C (Active Comparator): IUI 34-36 hours after HCG
  Interventions: Drug: HCG

INTERVENTIONS:
Drug: HCG — Women will be given HCG before IUI
  Other Names: Pregnyl

SUMMARY:
Evaluation of the effect of altering the timing of human chorionic gonadotropin (HCG) administration on the clinical pregnancy rate in intrauterine insemination (IUI) cycles.

DETAILED DESCRIPTION:
Women will be randomly divided into 3 groups; the first group will undergo IUI at the time HCG administration, the second group will undergo IUI 12 hours after HCG administration and the third group will undergo IUI 34-36 hours after HCG administration.

ELIGIBILITY:
Inclusion Criteria:

* Mild male factor infertility or unexplained infertility.

Exclusion Criteria:

* Advanced male factor infertility.
* Polycystic ovary syndrome (PCOS) as defined by the Rotterdam criteria.
* Endometriosis.
* Tubal disease.
* Uterine abnormalities or myoma.
* Previous uterine surgery.
* Metabolic or hormonal abnormalities.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4-6 weeks after IUI
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 4-6 weeks after IUI) divided by the number of IUI cycles

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Eid, Dr, Principal Investigator — Mansoura University
Locations (2):
- Egypt (2):
  - Fertility care unit (FCU) in Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate
  - Private fertility care centers, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: Undecided